CLINICAL TRIAL: NCT00138931
Title: Genetic Studies of Patients and Their Families With Inherited Cardiovascular and Neuromuscular Diseases.
Brief Title: Genetics of Cardiovascular and Neuromuscular Disease
Status: Recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 8249
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Cardiomyopathy; Arrhythmia; Muscular Dystrophy
Keywords: Cardiomyopathy; Arrhythmia; Muscular Dystrophy
MeSH Terms: conditions — Cardiomyopathies; Arrhythmias, Cardiac; Muscular Dystrophies | interventions — Blood Specimen Collection; Genetic Testing

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Blood draw (genetic testing) — Blood draw (genetic testing)

SUMMARY:
We are studying the genetics of human cardiovascular and neuromuscular disease. There are many different genetic regions that have been associated with the development of cardiomyopathy. An equal number of genetic regions have been associated with muscular dystrophy and there is overlap because some of the identical genes, when mutated, produce both cardiomyopathy and muscular dystrophy. We are working to identify genes and gene mutations associated with cardiomyopathy, arrhythmias and muscular dystrophy. We propose to screen these samples for mutations in genes known to be involved in these disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all ages will be considered for the study. In particular, families with more than one affected relative will be sought.

Exclusion Criteria:

* Subjects without a suspected inherited cardiovascular or neuromuscular disorder will be excluded from this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of all ages with familial idiopathic cardiomyopathy, including dilated, hypertrophic, and left ventricular non-compaction cardiomyopathy
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 1996-09; Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Identification of genetic causes of cardiomyopathy | unlimited

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth McNally, MD PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Noguchi S, McNally EM, Ben Othmane K, Hagiwara Y, Mizuno Y, Yoshida M, Yamamoto H, Bonnemann CG, Gussoni E, Denton PH, Kyriakides T, Middleton L, Hentati F, Ben Hamida M, Nonaka I, Vance JM, Kunkel LM, Ozawa E. Mutations in the dystrophin-associated protein gamma-sarcoglycan in chromosome 13 muscular dystrophy. Science. 1995 Nov 3;270(5237):819-22. doi: 10.1126/science.270.5237.819. PMID 7481775
- [Background] McNally EM, Duggan D, Gorospe JR, Bonnemann CG, Fanin M, Pegoraro E, Lidov HG, Noguchi S, Ozawa E, Finkel RS, Cruse RP, Angelini C, Kunkel LM, Hoffman EP. Mutations that disrupt the carboxyl-terminus of gamma-sarcoglycan cause muscular dystrophy. Hum Mol Genet. 1996 Nov;5(11):1841-7. doi: 10.1093/hmg/5.11.1841. PMID 8923014
- [Background] McNally EM, Passos-Bueno MR, Bonnemann CG, Vainzof M, de Sa Moreira E, Lidov HG, Othmane KB, Denton PH, Vance JM, Zatz M, Kunkel LM. Mild and severe muscular dystrophy caused by a single gamma-sarcoglycan mutation. Am J Hum Genet. 1996 Nov;59(5):1040-7. PMID 8900232
- [Background] van der Kooi AJ, van Meegen M, Ledderhof TM, McNally EM, de Visser M, Bolhuis PA. Genetic localization of a newly recognized autosomal dominant limb-girdle muscular dystrophy with cardiac involvement (LGMD1B) to chromosome 1q11-21. Am J Hum Genet. 1997 Apr;60(4):891-5. PMID 9106535
- [Background] Messina DN, Speer MC, Pericak-Vance MA, McNally EM. Linkage of familial dilated cardiomyopathy with conduction defect and muscular dystrophy to chromosome 6q23. Am J Hum Genet. 1997 Oct;61(4):909-17. doi: 10.1086/514896. PMID 9382102
- [Background] Davis DB, Delmonte AJ, Ly CT, McNally EM. Myoferlin, a candidate gene and potential modifier of muscular dystrophy. Hum Mol Genet. 2000 Jan 22;9(2):217-26. doi: 10.1093/hmg/9.2.217. PMID 10607832
- [Background] Nowak KJ, Walsh P, Jacob RL, Johnsen RD, Peverall J, McNally EM, Wilton SD, Kakulas BA, Laing NG. Severe gamma-sarcoglycanopathy caused by a novel missense mutation and a large deletion. Neuromuscul Disord. 2000 Feb;10(2):100-7. doi: 10.1016/s0960-8966(99)00063-2. PMID 10714584
- [Background] McNally EM, Ly CT, Rosenmann H, Mitrani Rosenbaum S, Jiang W, Anderson LV, Soffer D, Argov Z. Splicing mutation in dysferlin produces limb-girdle muscular dystrophy with inflammation. Am J Med Genet. 2000 Apr 10;91(4):305-12. doi: 10.1002/(sici)1096-8628(20000410)91:43.0.co;2-s. PMID 10766988
- [Background] de Paula F, Vainzof M, Bernardino AL, McNally E, Kunkel LM, Zatz M. Mutations in the caveolin-3 gene: When are they pathogenic? Am J Med Genet. 2001 Apr 1;99(4):303-7. doi: 10.1002/1096-8628(2001)9999:99993.0.co;2-o. PMID 11251997
- [Background] Vainzof M, Anderson LV, McNally EM, Davis DB, Faulkner G, Valle G, Moreira ES, Pavanello RC, Passos-Bueno MR, Zatz M. Dysferlin protein analysis in limb-girdle muscular dystrophies. J Mol Neurosci. 2001 Aug;17(1):71-80. doi: 10.1385/JMN:17:1:71. PMID 11665864
- [Background] McNally EM. Beta-myosin heavy chain gene mutations in familial hypertrophic cardiomyopathy: the usual suspect? Circ Res. 2002 Feb 22;90(3):246-7. No abstract available. PMID 11861410
- [Background] Wheeler MT, Zarnegar S, McNally EM. Zeta-sarcoglycan, a novel component of the sarcoglycan complex, is reduced in muscular dystrophy. Hum Mol Genet. 2002 Sep 1;11(18):2147-54. doi: 10.1093/hmg/11.18.2147. PMID 12189167
- [Background] McNally E, Allikian M, Wheeler MT, Mislow JM, Heydemann A. Cytoskeletal defects in cardiomyopathy. J Mol Cell Cardiol. 2003 Mar;35(3):231-41. doi: 10.1016/s0022-2828(03)00018-x. PMID 12676538
- [Background] MacLeod HM, Culley MR, Huber JM, McNally EM. Lamin A/C truncation in dilated cardiomyopathy with conduction disease. BMC Med Genet. 2003 Jul 10;4:4. doi: 10.1186/1471-2350-4-4. PMID 12854972
- [Background] Muchir A, van Engelen BG, Lammens M, Mislow JM, McNally E, Schwartz K, Bonne G. Nuclear envelope alterations in fibroblasts from LGMD1B patients carrying nonsense Y259X heterozygous or homozygous mutation in lamin A/C gene. Exp Cell Res. 2003 Dec 10;291(2):352-62. doi: 10.1016/j.yexcr.2003.07.002. PMID 14644157
- [Background] McNally EM, Towbin JA. Cardiomyopathy in muscular dystrophy workshop. 28-30 September 2003, Tucson, Arizona. Neuromuscul Disord. 2004 Jul;14(7):442-8. doi: 10.1016/j.nmd.2004.04.003. No abstract available. PMID 15266661
- [Background] DeWitt MM, MacLeod HM, Soliven B, McNally EM. Phospholamban R14 deletion results in late-onset, mild, hereditary dilated cardiomyopathy. J Am Coll Cardiol. 2006 Oct 3;48(7):1396-8. doi: 10.1016/j.jacc.2006.07.016. Epub 2006 Sep 12. PMID 17010801
- [Background] Heydemann A, Doherty KR, McNally EM. Genetic modifiers of muscular dystrophy: implications for therapy. Biochim Biophys Acta. 2007 Feb;1772(2):216-28. doi: 10.1016/j.bbadis.2006.06.013. Epub 2006 Jul 11. PMID 16916601
- [Background] Heydemann A, Demonbreun A, Hadhazy M, Earley JU, McNally EM. Nuclear sequestration of delta-sarcoglycan disrupts the nuclear localization of lamin A/C and emerin in cardiomyocytes. Hum Mol Genet. 2007 Feb 15;16(4):355-63. doi: 10.1093/hmg/ddl453. Epub 2006 Dec 12. PMID 17164264
- [Background] McNally EM. New approaches in the therapy of cardiomyopathy in muscular dystrophy. Annu Rev Med. 2007;58:75-88. doi: 10.1146/annurev.med.58.011706.144703. PMID 17217326
- [Background] Allikian MJ, McNally EM. Processing and assembly of the dystrophin glycoprotein complex. Traffic. 2007 Mar;8(3):177-83. doi: 10.1111/j.1600-0854.2006.00519.x. Epub 2007 Jan 26. PMID 17274800
- [Background] Heydemann A, McNally EM. Consequences of disrupting the dystrophin-sarcoglycan complex in cardiac and skeletal myopathy. Trends Cardiovasc Med. 2007 Feb;17(2):55-9. doi: 10.1016/j.tcm.2006.12.002. PMID 17292047
- [Background] McNally EM, Pytel P. Muscle diseases: the muscular dystrophies. Annu Rev Pathol. 2007;2:87-109. doi: 10.1146/annurev.pathol.2.010506.091936. PMID 18039094
- [Background] Dellefave L, McNally EM. Sarcomere mutations in cardiomyopathy, noncompaction, and the developing heart. Circulation. 2008 Jun 3;117(22):2847-9. doi: 10.1161/CIRCULATIONAHA.108.781518. No abstract available. PMID 18519860
- [Background] MacLeod HM, McNally EM. A pilot study of a family history risk assessment tool for cardiovascular disease. J Genet Couns. 2008 Oct;17(5):499-507. doi: 10.1007/s10897-008-9174-z. Epub 2008 Sep 13. PMID 18791812
- [Background] Puckelwartz MJ, Kessler EJ, Kim G, Dewitt MM, Zhang Y, Earley JU, Depreux FF, Holaska J, Mewborn SK, Pytel P, McNally EM. Nesprin-1 mutations in human and murine cardiomyopathy. J Mol Cell Cardiol. 2010 Apr;48(4):600-8. doi: 10.1016/j.yjmcc.2009.11.006. Epub 2009 Nov 24. PMID 19944109
- [Background] Dellefave L, McNally EM. The genetics of dilated cardiomyopathy. Curr Opin Cardiol. 2010 May;25(3):198-204. doi: 10.1097/HCO.0b013e328337ba52. PMID 20186049
- [Background] Romfh A, McNally EM. Cardiac assessment in duchenne and becker muscular dystrophies. Curr Heart Fail Rep. 2010 Dec;7(4):212-8. doi: 10.1007/s11897-010-0028-2. PMID 20857240
- [Background] Swaggart KA, Heydemann A, Palmer AA, McNally EM. Distinct genetic regions modify specific muscle groups in muscular dystrophy. Physiol Genomics. 2011 Jan 7;43(1):24-31. doi: 10.1152/physiolgenomics.00172.2010. Epub 2010 Oct 19. PMID 20959497
- [Background] McNally EM, Patel AR. Cardiac magnetic resonance of left ventricular trabeculation: the new normal. Circ Cardiovasc Imaging. 2011 Mar;4(2):84-6. doi: 10.1161/CIRCIMAGING.110.962472. No abstract available. PMID 21406661
- [Background] Posey AD Jr, Demonbreun A, McNally EM. Ferlin proteins in myoblast fusion and muscle growth. Curr Top Dev Biol. 2011;96:203-30. doi: 10.1016/B978-0-12-385940-2.00008-5. PMID 21621072
- [Background] McNally EM, Sparano D. Mechanisms and management of the heart in myotonic dystrophy. Heart. 2011 Jul;97(13):1094-100. doi: 10.1136/hrt.2010.214197. PMID 21642660
- [Background] Puckelwartz MJ, Depreux FF, McNally EM. Gene expression, chromosome position and lamin A/C mutations. Nucleus. 2011 May-Jun;2(3):162-7. doi: 10.4161/nucl.2.3.16003. PMID 21818408
- [Background] Golbus JR, Puckelwartz MJ, Fahrenbach JP, Dellefave-Castillo LM, Wolfgeher D, McNally EM. Population-based variation in cardiomyopathy genes. Circ Cardiovasc Genet. 2012 Aug 1;5(4):391-9. doi: 10.1161/CIRCGENETICS.112.962928. Epub 2012 Jul 4. PMID 22763267
- [Background] Flanigan KM, Ceco E, Lamar KM, Kaminoh Y, Dunn DM, Mendell JR, King WM, Pestronk A, Florence JM, Mathews KD, Finkel RS, Swoboda KJ, Gappmaier E, Howard MT, Day JW, McDonald C, McNally EM, Weiss RB; United Dystrophinopathy Project. LTBP4 genotype predicts age of ambulatory loss in Duchenne muscular dystrophy. Ann Neurol. 2013 Apr;73(4):481-8. doi: 10.1002/ana.23819. Epub 2013 Feb 20. PMID 23440719
- [Result] MacLeod H, Pytel P, Wollmann R, Chelmicka-Schorr E, Silver K, Anderson RB, Waggoner D, McNally EM. A novel FKRP mutation in congenital muscular dystrophy disrupts the dystrophin glycoprotein complex. Neuromuscul Disord. 2007 Apr;17(4):285-9. doi: 10.1016/j.nmd.2007.01.005. Epub 2007 Mar 1. PMID 17336067
- [Result] Lakdawala NK, Dellefave L, Redwood CS, Sparks E, Cirino AL, Depalma S, Colan SD, Funke B, Zimmerman RS, Robinson P, Watkins H, Seidman CE, Seidman JG, McNally EM, Ho CY. Familial dilated cardiomyopathy caused by an alpha-tropomyosin mutation: the distinctive natural history of sarcomeric dilated cardiomyopathy. J Am Coll Cardiol. 2010 Jan 26;55(4):320-9. doi: 10.1016/j.jacc.2009.11.017. PMID 20117437
- [Result] Puckelwartz MJ, Pesce LL, Nelakuditi V, Dellefave-Castillo L, Golbus JR, Day SM, Cappola TP, Dorn GW 2nd, Foster IT, McNally EM. Supercomputing for the parallelization of whole genome analysis. Bioinformatics. 2014 Jun 1;30(11):1508-13. doi: 10.1093/bioinformatics/btu071. Epub 2014 Feb 12. PMID 24526712
- [Derived] Dellefave LM, Pytel P, Mewborn S, Mora B, Guris DL, Fedson S, Waggoner D, Moskowitz I, McNally EM. Sarcomere mutations in cardiomyopathy with left ventricular hypertrabeculation. Circ Cardiovasc Genet. 2009 Oct;2(5):442-9. doi: 10.1161/CIRCGENETICS.109.861955. Epub 2009 Jul 24. PMID 20031619